CLINICAL TRIAL: NCT03515395
Title: Acceptance and Frequency of Use of a Computer Game Based Exercise Training in Geriatric Patients After Hip Fracture Surgery
Brief Title: Entertainement and Training After a Hip Fracture
Acronym: ENTERAIN-HF
Status: Withdrawn | Type: Observational
Why Stopped: Low recruitement, no scientific staff
Sponsor: Geriatrische Klinik St. Gallen (Other)
Responsible Party: Principal Investigator, Thomas Munzer, MD, PhD, Head Department of Geriatrics, Geriatrische Klinik St. Gallen
Other Study IDs: BASEC 2018-00528
Record Dates: First submitted 2018-04-19; First posted 2018-05-03 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2019-05

CONDITIONS: Hip Fractures; Exercise; Aging
Keywords: exergaming; hip fracture; training; acceptance
MeSH Terms: conditions — Hip Fractures; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Instruction to a computer game and motivation to use it — Patients who are willing to use the computer game and who have given written informed consent shall have three instruction sessions by a physiotherapist instructor. They will then asked to use the platform at least 3 times per week at their own discretion. The platform will be installed in the patient room, alternatively in a defined training room. The patient will be free to choose the time and duration of the gaming. This allows the patients to select times that do not interfere with their usual therapy schedule or visits (e.g. evening or weekends). Prior to discharge compliance with the platform will be monitored by analyzing the gaming data of each patient.

SUMMARY:
Older persons are at riskt for falls and fractures. After hip surgery they are normally treated with physical or occupational therapy. The additional use of computer based exercise games for training and the acceptance of such a technology are unclear. Thus, we plant to assess the above outcome ins an observational pilot study.

DETAILED DESCRIPTION:
Falls and fall-associated fractures have a big medical burden on our societies. Older persons who suffer from a fall that leads to a trauma and fracture often loose functional capacity. They may have prolonged mobility problems and are at risk for long-term care or nursing home institutionalization. To date, measures to prevent such negative outcomes are early mobilization and functional physical or occupational therapy immediately following orthopedic surgery. In addition, patients usually are asked to train at home after hospital discharge. This can be achieved by a home training program or by ambulatory physical therapy. Recent technological development has introduced computerized training and gaming platforms into geriatric rehabilitation settings and home exercise training. Games that have been developed for a younger population have now been adapted to the needs of older persons. A recent systematic review has demonstrated that such platforms. for example Wii significantly improve balance and therefore have the potential to prevent falls]. However to date such platforms have not been evaluated in a defined geriatric hospital patient population (e.g. after a hip fracture) as an adjunct to in-hospital physical therapy. Thus, such platforms could be offered as an additional training opportunity.

ELIGIBILITY:
Inclusion Criteria:

Living at home or in a retirement home (independent living situation) Time between surgery and the start of the gaming intervention less or equal 10 days Patient must be able to ambulate and to have full weight bearing

Exclusion Criteria:

The following exclusion criteria will apply

* Acute delirium (daily delirium observation score > 3 during the first three consecutive days) lasting for more than 10 days. If the delirium resolves within the 10 day period (see above) patients without cognitive decline are still eligible.
* A history of severe dementia prior to admission or poor cognition at admission after exclusion of delirium (MOCA score < 15 or MMT < 15).
* Patients who were initially admitted from a nursing home

Ages: 75 Years to 105 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients age 75 and older who sufferd from a trauma leading to a hip fracture Surgical procedure: intramedullary gamma nail osteosynthesis (IGNOS, gamma nail)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptance of technology | 14 days of game use
  Questionnaire based answers about computer game use

SECONDARY OUTCOMES:
Functional improvement | after 14 days of game use
  Measurement of mobility (short physical performance battery test) score hand grip strength in both hands (kPa) the best of three trials will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Münzer, MD, Principal Investigator — Geriatrische Klinik St. Gallen
Locations (1):
- Geriatrische Klinik, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Sharing depends of the quality of the collected data

REFERENCES:
- [Background] Tinetti ME, Williams CS. The effect of falls and fall injuries on functioning in community-dwelling older persons. J Gerontol A Biol Sci Med Sci. 1998 Mar;53(2):M112-9. doi: 10.1093/gerona/53a.2.m112. PMID 9520917
- [Background] Campbell AJ, Reinken J, Allan BC, Martinez GS. Falls in old age: a study of frequency and related clinical factors. Age Ageing. 1981 Nov;10(4):264-70. doi: 10.1093/ageing/10.4.264. PMID 7337066
- [Background] Karahan AY, Tok F, Taskin H, Kucuksarac S, Basaran A, Yildirim P. Effects of Exergames on Balance, Functional Mobility, and Quality of Life of Geriatrics Versus Home Exercise Programme: Randomized Controlled Study. Cent Eur J Public Health. 2015 Nov;23 Suppl:S14-8. doi: 10.21101/cejph.a4081. PMID 26849537
- [Background] van Diest M, Lamoth CJ, Stegenga J, Verkerke GJ, Postema K. Exergaming for balance training of elderly: state of the art and future developments. J Neuroeng Rehabil. 2013 Sep 25;10:101. doi: 10.1186/1743-0003-10-101. PMID 24063521
- [Result] Chao YY, Scherer YK, Montgomery CA. Effects of using Nintendo Wii exergames in older adults: a review of the literature. J Aging Health. 2015 Apr;27(3):379-402. doi: 10.1177/0898264314551171. Epub 2014 Sep 21. PMID 25245519